CLINICAL TRIAL: NCT01696032
Title: A Randomized, Controlled, Open-Label, Phase 2 Trial of SGI-110 and Carboplatin in Subjects With Platinum-Resistant Recurrent Ovarian Cancer
Brief Title: SGI-110 in Combination With Carboplatin in Ovarian Cancer
Acronym: SGI-110
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGI-110-02
Record Dates: First submitted 2012-09-26; First posted 2012-09-28 (Estimated); Results first posted 2021-05-25 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-07

CONDITIONS: Ovarian Cancer
Keywords: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — guadecitabine; Topotecan; liposomal doxorubicin; Paclitaxel; Gemcitabine; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SGI-110 + Carboplatin (Experimental): Stage 1 was a safety lead-in stage with a dose escalation design. Participants were evaluated with the combination of SGI-110 (guadecitabine) plus carboplatin (G+C), given as 28-day treatment cycles: guadecitabine administered subcutaneous (SC) daily on Days 1-5, at a starting dose of 45 mg/m2/day in Cohort 1, followed by carboplatin intravenous (IV) based on a targeted dose of area under the curve (AUC) 5 on Day 8. After dose limiting toxicities were noted, guadecitabine dose was reduced to 30 mg/m2/day for subsequent cycles for 4 participants. Cohort 2 received 30 mg/m2/day guadecitabine and carboplatin IV AUC 4.
  Interventions: Drug: SGI-110; Drug: Carboplatin
- SGI-110 + Carboplatin or TC (Experimental): Stage 2 was an open-label, randomized, controlled trial. Eligible participants were randomly assigned in a 1:1 ratio to receive either (1) G+C combination treatment in 28-day cycles at 30 mg/m2 SC once daily on Days 1-5 and carboplatin IV AUC 4 on Day 8, or (2) treatment of choice (TC) of topotecan, pegylated liposomal doxorubicin (PLD), paclitaxel, or gemcitabine based on recommended dosing in 28-day cycles; participants initially randomized to TC were able to cross over to receive 30 mg/m2 G+C due to disease progression.
  Interventions: Drug: SGI-110; Drug: Treatment of Choice (topotecan, pegylated liposomal doxorubicin, paclitaxel, or gemcitabine); Drug: Carboplatin

INTERVENTIONS:
Drug: SGI-110
  Other Names: guadecitabine
Drug: Treatment of Choice (topotecan, pegylated liposomal doxorubicin, paclitaxel, or gemcitabine) — Investigator chose to treat with either topotecan, pegylated liposomal doxorubicin, paclitaxel, or gemcitabine
  Arms: SGI-110 + Carboplatin or TC
Drug: Carboplatin

SUMMARY:
A 2-part, Phase 2 controlled, open-label, randomized study in participants with platinum-resistant recurrent ovarian cancer. In Part 1, participants received SGI-110 and carboplatin. The optimum dose of SGI-110 (guadecitabine) was identified in Part 1 based on safety and efficacy. In Part 2, participants were randomized to receive the dose identified in Part 1 plus carboplatin or one of four treatment of choice at the discretion of the investigator. The treatment of choice consisted of topotecan, pegylated liposomal doxorubicin, paclitaxel or gemcitabine.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who are women 18 years of age or older.
2. Participants who have histologically or cytologically confirmed recurrent high-grade serous epithelial ovarian cancer (Grade 2 or 3), primary peritoneal carcinomatosis or fallopian tube cancer.
3. Participants who have platinum-resistant disease (defined as having relapsed within 6 months of her last platinum-containing regimen). There is no limit on the number of prior treatment regimens in Part 1. In Part 2, participants may have had no more than 3 prior cytotoxic treatment regimens, excluding adjuvant or maintenance therapy.
4. Participants must have had prior paclitaxel treatment.
5. Participants who have measurable disease according to RECIST v1.1 or detectable disease.
6. Participants with ECOG performance status of 0 or 1.
7. Participants with acceptable organ function.
8. Participants must be at least 3 weeks from last chemotherapy.

Exclusion Criteria:

1. Participants who have hypersensitivity to SGI-110 and/or carboplatin or other components of these drug products.
2. Participants who have received prior therapy with any hypomethylating agents.
3. Participants who are refractory to platinum treatment i.e., progressed while on platinum treatment.
4. Participants with abnormal left ventricular ejection fraction.
5. Participants with Grade 2 or greater neuropathy.
6. Participants with known brain metastases.
7. Participants with known history of HIV, HCV or HBV.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-09; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (24):
- United States (13):
  - Norris Comprehensive Cancer Center- University of Southern California, Los Angeles, California
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Georgia Health Sciences University, Augusta, Georgia
  - University of Chicago, Chicago, Illinois
  - Melvin and Bren Simon Cancer Center- Indiana University, Indianapolis, Indiana
  - Women's Cancer Care, Covington, Louisiana
  - Johns Hopkins Kimmel Cancer Center, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Island Gynecologic Oncology, Brightwaters, New York
  - Duke Cancer Institute- Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati Cancer Institute, Cincinnati, Ohio
  - Mary Crowley Medical Research Center, Dallas, Texas
  - Inova Fairfax Hospital, Falls Church, Virginia
- Canada (4):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - CHUM Gynecologie-Oncologie, Notre Dame Hospital, Montreal, Quebec
- United Kingdom (7):
  - Bristol Heamatology and Oncology Centre, Bristol
  - St. James Univesity Hospital - St. James Institute of Oncology, Leeds
  - Cambridge University Hospitals NHS Foundation and Trust, London
  - Univesity College Hospital, London
  - Imperial College Health Care NHS Trust-Garry Weston Centre, London
  - Mount Vernon Cancer Centre, Middlesex
  - Royal Marsden Foundation Trust, Sutton

REFERENCES:
- [Derived] Cardenas H, Fang F, Jiang G, Perkins SM, Zhang C, Emerson RE, Hutchins G, Keer HN, Liu Y, Matei D, Nephew K. Methylomic Signatures of High Grade Serous Ovarian Cancer. Epigenetics. 2021 Nov;16(11):1201-1216. doi: 10.1080/15592294.2020.1853402. Epub 2020 Dec 8. PMID 33289590
- [Derived] Oza AM, Matulonis UA, Alvarez Secord A, Nemunaitis J, Roman LD, Blagden SP, Banerjee S, McGuire WP, Ghamande S, Birrer MJ, Fleming GF, Markham MJ, Hirte HW, Provencher DM, Basu B, Kristeleit R, Armstrong DK, Schwartz B, Braly P, Hall GD, Nephew KP, Jueliger S, Oganesian A, Naim S, Hao Y, Keer H, Azab M, Matei D. A Randomized Phase II Trial of Epigenetic Priming with Guadecitabine and Carboplatin in Platinum-resistant, Recurrent Ovarian Cancer. Clin Cancer Res. 2020 Mar 1;26(5):1009-1016. doi: 10.1158/1078-0432.CCR-19-1638. Epub 2019 Dec 12. PMID 31831561

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 124 participants were enrolled in the study and 120 were treated at 20 study centers, with 12 in the United States, 5 in the United Kingdom, and 3 in Canada. The enrollment period was 10 December 2012 (first participant dosed) to 12 May 2014 (last participant first dose).
Groups:
- Stage 1: Guadecitabine+Carboplatin 30 mg/m2; Stage 2: Guadecitabine+Carboplatin 30 mg/m2: Guadecitabine 30 mg/m2 on Days 1-5 and carboplatin AUC 4 on Day 8 of 28-day treatment cycles.
- Stage 1: Guadecitabine+Carboplatin 45 mg/m2: Guadecitabine 45 mg/m2 on Days 1-5 and carboplatin AUC 4 on Day 8 of 28-day treatment cycles. Due to dose limiting toxicities, the guadecitabine dose for this group was reduced from 45 mg/m2 to 30 mg/m2 after Cycle 1 for 4 of 6 participants and the carboplatin dose was reduced for 2 of 6 participants.
- Stage 2: Treatment Choice: Treatment was selected at the investigator's discretion and administered based on recommended dosing for topotecan (3.5-4.0 mg/m2/wk administered on Days 1, 8, and 15 via IV infusion); pegylated liposomal doxorubicin (PLD) (40-50 mg/m2 administered on Day 1 via IV infusion), paclitaxel (60-80 mg/m2/wk administered on Days 1, 8, 15, and 22 via IV infusion), or gemcitabine (800-1000 mg/m2 administered on Days 1, 8, and 15 via IV infusion). Participants initially randomized to TC were able to cross over to receive 30 mg/m2 G+C due to disease progression.
Period: Overall Study
Arm/Group | Stage 1: Guadecitabine+Carboplatin 30 mg/m2 | Stage 1: Guadecitabine+Carboplatin 45 mg/m2 | Stage 2: Guadecitabine+Carboplatin 30 mg/m2 | Stage 2: Treatment Choice
Started | 14 | 6 | 51 | 49
Completed | 0 | 0 | 0 | 27
Not Completed | 14 | 6 | 51 | 22
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 2
Not completed — Death | 14 | 4 | 43 | 18
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Database lock | 0 | 1 | 7 | 2

BASELINE CHARACTERISTICS:
Population: Includes all treated participants
Groups:
- Stage 2: Treatment Choice: Treatment was selected at the investigator's discretion and administered based on recommended dosing for topotecan (3.5-4.0 mg/m2/wk administered on Days 1, 8, and 15 via IV infusion); PLD (40-50 mg/m2 administered on Day 1 via IV infusion), paclitaxel (60-80 mg/m2/wk administered on Days 1, 8, 15, and 22 via IV infusion), or gemcitabine (800-1000 mg/m2 administered on Days 1, 8, and 15 via IV infusion. Participants initially randomized to TC were able to cross over to receive 30 mg/m2 G+C due to disease progression.
- Total: Total of all reporting groups
Arm/Group | Stage 1: Guadecitabine+Carboplatin 30 mg/m2 | Stage 1: Guadecitabine+Carboplatin 45 mg/m2 | Stage 2: Guadecitabine+Carboplatin 30 mg/m2 | Stage 2: Treatment Choice | Total
Number analyzed (Participants) | 14 | 6 | 51 | 49 | 120
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.99 (9.47) | 56.79 (13.20) | 61.96 (9.17) | 62.09 (9.62) | 61.29 (9.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 6 | 51 | 49 | 120
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 2 | 3 | 6
  Not Hispanic or Latino | 13 | 6 | 49 | 46 | 114
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 5 | 5 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1
  Black or African American | 1 | 0 | 2 | 2 | 5
  White | 12 | 5 | 43 | 40 | 100
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Stage 1: Dose Limiting Toxicities
Description: Number of participants with dose limiting toxicities (DLTs) in Stage 1
Time Frame: Up to 12 months
Population: Safety data set includes data from all participants who received any amount of study drug, including any component of a multi-dose study treatment regimen.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1: Guadecitabine+Carboplatin 30 mg/m2 | Stage 1: Guadecitabine+Carboplatin 45 mg/m2
Number analyzed (Participants) | 14 | 6
Participants | 0 | 4

2. Primary Outcome: Stage 2: Progression Free Survival
Description: Progression free survival (PFS) time was defined as the time interval from the date of the first dose of study medication until the earlier of disease progression or death. Participants were treated with their assigned treatment [guadecitabine+carboplatin (G+C) or treatment choice (TC)] until disease progression or unacceptable treatment-related toxicity occurred.
Time Frame: Up to 24 months
Population: Efficacy data set included all participants who received any amount of study drug.
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- Stage 2: Treatment Choice: Treatment was selected at the investigator's discretion and administered based on recommended dosing for topotecan (3.5-4.0 mg/m2/wk administered on Days 1, 8, and 15 via IV infusion); PLD (40-50 mg/m2 administered on Day 1 via IV infusion), paclitaxel (60-80 mg/m2/wk administered on Days 1, 8, 15, and 22 via IV infusion), or gemcitabine (800-1000 mg/m2 administered on Days 1, 8, and 15 via IV infusion).
Arm/Group | Stage 2: Guadecitabine+Carboplatin 30 mg/m2 | Stage 2: Treatment Choice
Number analyzed (Participants) | 51 | 49
Days | 114 [63 to 169] | 64 [52 to 105]
Statistical Analysis 1: Comparison: Stage 2: Guadecitabine+Carboplatin 30 mg/m2 vs Stage 2: Treatment Choice; Test type: Superiority; p = 0.0654, Log Rank

3. Secondary Outcome: Objective Response Rate
Description: The objective response rate (ORR) was defined as the proportion of participants who experienced an objective response (best overall response of complete response/full response or partial response, which was confirmed by a subsequent assessment at least 28 days later). Response categories were determined based on RECIST v1.1 criteria, or on modified Rustin (CA-125) criteria if response assessment could not be made using RECIST criteria.
Time Frame: Up to 24 months
Population: Efficacy data set included all participants who received any amount of study drug.
Measure: Number (95% Confidence Interval); unit: Percent
Groups:
- Stage 2: Crossover Treatment Choice to Guadecitabine+Carboplatin 30 mg/m2: Crossover from treatment choice to the guadecitabine+carboplatin combination treatment arm was permitted for participants after evidence of disease progression.
Arm/Group | Stage 1: Guadecitabine+Carboplatin 30 mg/m2 | Stage 1: Guadecitabine+Carboplatin 45 mg/m2 | Stage 2: Guadecitabine+Carboplatin 30 mg/m2 | Stage 2: Treatment Choice | Stage 2: Crossover Treatment Choice to Guadecitabine+Carboplatin 30 mg/m2
Number analyzed (Participants) | 14 | 6 | 51 | 49 | 27
Percent | 21 [4.7 to 50.8] | 0 [0.0 to 45.9] | 16 [7.0 to 28.6] | 8 [2.3 to 19.6] | 4 [0.1 to 19.0]

4. Secondary Outcome: Progression Free Survival at 6 Months
Description: Progression free survival rate at 6 months is the proportion of participants who were alive and did not have disease progression at 6 months after start of treatment.
Time Frame: 6 months
Population: Efficacy data set included all participants who received any amount of study drug.
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Stage 1: Guadecitabine+Carboplatin 30 mg/m2 | Stage 1: Guadecitabine+Carboplatin 45 mg/m2 | Stage 2: Guadecitabine+Carboplatin 30 mg/m2 | Stage 2: Treatment Choice | Stage 2: Crossover Treatment Choice to Guadecitabine+Carboplatin 30 mg/m2
Number analyzed (Participants) | 14 | 6 | 51 | 49 | 27
Percent of participants | 0.36 [0.13 to 0.59] | 0.33 [0.05 to 0.68] | 0.37 [0.24 to 0.50] | 0.11 [0.04 to 0.22] | 0.19 [0.07 to 0.35]

5. Secondary Outcome: Clinical Benefit Rate
Description: Clinical benefit rate (CBR) was defined as the proportion of subjects who experienced a best overall response of complete response/full response or partial response (confirmed by a subsequent assessment at least 28 days later), or documented stable disease for at least 3 months after the first dose. Response categories were determined based on RECIST v1.1 criteria, then based on modified Rustin (CA-125) criteria if assessment could not be made using RECIST criteria.
Time Frame: Up to 24 months
Population: Efficacy data set included all participants who received any amount of study drug.
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Stage 1: Guadecitabine+Carboplatin 30 mg/m2 | Stage 1: Guadecitabine+Carboplatin 45 mg/m2 | Stage 2: Guadecitabine+Carboplatin 30 mg/m2 | Stage 2: Treatment Choice | Stage 2: Crossover Treatment Choice to Guadecitabine+Carboplatin 30 mg/m2
Number analyzed (Participants) | 14 | 6 | 51 | 49 | 27
Percent of participants | 43 [17.7 to 71.1] | 50 [11.8 to 88.2] | 41 [27.6 to 55.8] | 29 [16.6 to 43.3] | 19 [6.3 to 38.1]

6. Secondary Outcome: CA-125 Levels
Description: Percentage of participants with CA-125 reduction by ≥ 50% from baseline
Time Frame: Up to 24 months
Population: Efficacy data set included all participants who received any amount of study drug.
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Stage 1: Guadecitabine+Carboplatin 30 mg/m2 | Stage 1: Guadecitabine+Carboplatin 45 mg/m2 | Stage 2: Guadecitabine+Carboplatin 30 mg/m2 | Stage 2: Treatment Choice | Stage 2: Crossover Treatment Choice to Guadecitabine+Carboplatin 30 mg/m2
Number analyzed (Participants) | 14 | 6 | 51 | 49 | 27
Percent of participants | 27 [6.0 to 61.0] | 50 [6.8 to 93.2] | 36 [21.6 to 52.0] | 32 [18.1 to 48.1] | 29 [11.3 to 52.2]

7. Secondary Outcome: Duration of Response
Description: Duration of response is defined as the time between the date of the first documentation of complete response/full response or partial response, and the date of disease progression or date of death due to any cause, or the last adequate tumor assessment prior to the start of subsequent anti-cancer therapy including crossing over to G+C from TC arm, whichever occurred earlier. Only participants who responded were included in the duration of response calculation.
Time Frame: Up to 24 months
Population: Efficacy data set included all participants who received any amount of study drug.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Stage 1: Guadecitabine+Carboplatin 30 mg/m2 | Stage 1: Guadecitabine+Carboplatin 45 mg/m2 | Stage 2: Guadecitabine+Carboplatin 30 mg/m2 | Stage 2: Treatment Choice | Stage 2: Crossover Treatment Choice to Guadecitabine+Carboplatin 30 mg/m2
Number analyzed (Participants) | 6 | 3 | 21 | 14 | 5
Days | 225 [42.0 to 294.0] | 195 [114.0 to NA] — Not estimable with current data | 186 [147.0 to 241.0] | 173 [121.0 to 267.0] | 182 [147.0 to 233.0]

8. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the number of days from the day the participant was administered the first dose of study treatment to the date of death (regardless of cause). Survival time was censored on the last date the participant was known to be alive or lost to follow-up before reaching the event of death; in the TC group, time was censored at the date of crossover.
Time Frame: Up to 24 months
Population: Efficacy data set included all participants who received any amount of study drug.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Stage 1: Guadecitabine+Carboplatin 30 mg/m2 | Stage 1: Guadecitabine+Carboplatin 45 mg/m2 | Stage 2: Guadecitabine+Carboplatin 30 mg/m2 | Stage 2: Treatment Choice | Stage 2: Crossover Treatment Choice to Guadecitabine+Carboplatin 30 mg/m2
Number analyzed (Participants) | 14 | 6 | 51 | 49 | 27
Days | 341 [100.0 to 567.0] | 195 [25.0 to NA] — Not estimable with current data | 331 [231 to 415] | 221 [145 to 372] | 279 [161.0 to 413.0]

9. Secondary Outcome: Stage 1: Pharmacokinetic Parameter Cmax
Description: Time to maximum plasma concentration for guadecitabine, decitabine and carboplatin
Time Frame: Pre-dose and up to 8 hours post-dose on Cycle 1 Day 1 for guadecitabine and decitabine and Day 8 for carboplatin (28 day cycles)
Population: The pharmacokinetic (PK) population included participants for which sufficient data were available to calculate PK parameters.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Stage 1: Guadecitabine+Carboplatin 30 mg/m2 | Stage 1: Guadecitabine+Carboplatin 45 mg/m2
Number analyzed (Participants) | 14 | 5
ng/mL
  Guadecitabine | 96.2 (78.3) | 109 (70.8)
  Decitabine | 22.6 (13.3) | 26.3 (14.5)
  Carboplatin | 19600 (5650) | 21900 (13800)

10. Secondary Outcome: Stage 1: Pharmacokinetic Parameter Tmax
Description: Time to last measurable concentration for guadecitabine, decitabine and carboplatin
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Median (Full Range); unit: Hours
Arm/Group | Stage 1: Guadecitabine+Carboplatin 30 mg/m2 | Stage 1: Guadecitabine+Carboplatin 45 mg/m2
Number analyzed (Participants) | 14 | 5
Hours
  Guadecitabine | 1.42 [0.25 to 6.00] | 1.98 [1.50 to 7.25]
  Decitabine | 1.98 [1.00 to 6.00] | 3.95 [1.67 to 7.25]
  Carboplatin | 1.03 [0.48 to 1.20] | 1.05 [0.48 to 1.20]

11. Secondary Outcome: Stage 1: Pharmacokinetic Parameter AUC0-8
Description: Area under the concentration-time curve from 0 to 8 hours (AUC0-8) for guadecitabine, decitabine and carboplatin
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Hours*ng/mL
Arm/Group | Stage 1: Guadecitabine+Carboplatin 30 mg/m2 | Stage 1: Guadecitabine+Carboplatin 45 mg/m2
Number analyzed (Participants) | 13 | 4
Hours*ng/mL
  Guadecitabine | 239 (136) | 416 (217)
  Decitabine | 71.1 (26.6) | 129 (17.9)
  Carboplatin | 51200 (12100) | 41900 (31700)

ADVERSE EVENTS:
Time Frame: Approximately 4 years
Description: Treatment-emergent adverse events (TEAEs) were defined as events that first occurred or worsened after the first dose of study drug given on Cycle 1 Day 1 until 30 days after the last dose of study treatment.
Arm/Group | Stage 1: Guadecitabine+Carboplatin 30 mg/m2 | Stage 1: Guadecitabine+Carboplatin 45 mg/m2 | Stage 2: Guadecitabine+Carboplatin 30 mg/m2 | Stage 2: Treatment Choice | Stage 2: Crossover Treatment Choice to Guadecitabine+Carboplatin 30 mg/m2
All-Cause Mortality (participants affected / at risk) | 14/14 | 4/6 | 43/51 | 18/49 | 22/27
Serious Adverse Events (participants affected / at risk) | 8/14 | 4/6 | 26/51 | 24/49 | 12/27
Other Adverse Events (participants affected / at risk) | 14/14 | 6/6 | 50/51 | 49/49 | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage 1: Guadecitabine+Carboplatin 30 mg/m2 (N=14) | Stage 1: Guadecitabine+Carboplatin 45 mg/m2 (N=6) | Stage 2: Guadecitabine+Carboplatin 30 mg/m2 (N=51) | Stage 2: Treatment Choice (N=49) | Stage 2: Crossover Treatment Choice to Guadecitabine+Carboplatin 30 mg/m2 (N=27)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Adverse drug reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Elective procedure (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mental status change (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
International normalized ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (3) | 3 (3) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral neuropathy sensory (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Radicular pain (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0) | 8 (8) | 4 (4) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 5 (5)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 5 (5) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4) | 4 (4) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal abscess (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gait disturbance (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infections (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Postoperative fever (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage 1: Guadecitabine+Carboplatin 30 mg/m2 (N=14) | Stage 1: Guadecitabine+Carboplatin 45 mg/m2 (N=6) | Stage 2: Guadecitabine+Carboplatin 30 mg/m2 (N=51) | Stage 2: Treatment Choice (N=49) | Stage 2: Crossover Treatment Choice to Guadecitabine+Carboplatin 30 mg/m2 (N=27)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 7 (7) | 6 (6) | 2 (2)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Flushing (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 3 (3)
Lymphedema (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Fatigue (General disorders) | 9 (9) | 4 (4) | 33 (33) | 26 (26) | 14 (14)
Injection site reaction (General disorders) | 8 (8) | 2 (2) | 23 (23) | 1 (1) | 9 (9)
Pyrexia (General disorders) | 2 (2) | 4 (4) | 8 (8) | 3 (3) | 3 (3)
Peripheral edema (General disorders) | 2 (2) | 2 (2) | 5 (5) | 14 (14) | 3 (3)
Adverse drug reaction (General disorders) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 4 (4)
Pain (General disorders) | 0 (0) | 0 (0) | 5 (5) | 4 (4) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 1 (1)
Hernia pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Early satiety (General disorders) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Injection site pain (General disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mass (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 3 (3) | 2 (2) | 6 (6) | 6 (6) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 4 (4) | 13 (13) | 3 (3)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 4 (4) | 5 (5) | 0 (0)
Libido decreased (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Perineal pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Vaginal ulceration (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal swelling (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 5 (5) | 1 (1) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 3 (3)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 3 (3) | 0 (0) | 2 (2)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Stoma site pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 2 (2) | 5 (5) | 0 (0)
Anion gap increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase (Investigations) | 2 (2) | 0 (0) | 4 (4) | 2 (2) | 2 (2)
Bilirubin urine present (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood albumin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 2 (2) | 0 (0) | 2 (2) | 4 (4) | 1 (1)
Blood chloride decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carbon dioxide decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Protein urine present (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (1) | 3 (3) | 2 (2) | 2 (2)
Specific gravity urine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine ketone body present (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine leukocyte esterase positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood phosphorous decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Protein total decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 7 (7) | 3 (3) | 2 (2)
International normalized ratio increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 7 (7) | 5 (5) | 36 (36) | 16 (16) | 18 (18)
Leukopenia (Blood and lymphatic system disorders) | 5 (5) | 2 (2) | 16 (16) | 11 (11) | 12 (12)
Anemia (Blood and lymphatic system disorders) | 7 (7) | 4 (4) | 16 (16) | 25 (25) | 8 (8)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 6 (6) | 12 (12) | 12 (12) | 10 (10)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 14 (14) | 15 (15) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 7 (7) | 8 (8) | 4 (4)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (3) | 3 (3) | 0 (0)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 5 (5) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 0 (0) | 9 (9) | 5 (5) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 5 (5) | 6 (6) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 4 (4) | 0 (0)
Parasthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 10 (10) | 2 (2) | 38 (38) | 28 (28) | 12 (12)
Vomiting (Gastrointestinal disorders) | 6 (6) | 2 (2) | 32 (32) | 15 (15) | 10 (10)
Constipation (Gastrointestinal disorders) | 5 (5) | 4 (4) | 22 (22) | 17 (17) | 10 (10)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 2 (2) | 21 (21) | 17 (17) | 8 (8)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 1 (1) | 21 (21) | 11 (11) | 9 (9)
Stomatitis (Gastrointestinal disorders) | 3 (3) | 1 (1) | 11 (11) | 12 (12) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 10 (10) | 12 (12) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 2 (2) | 6 (6) | 10 (10) | 3 (3)
Ascites (Gastrointestinal disorders) | 2 (2) | 2 (2) | 4 (4) | 4 (4) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 2 (2) | 8 (8) | 4 (4) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 0 (0) | 4 (4) | 5 (5) | 3 (3)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 3 (3)
Anorectal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 4 (4) | 2 (2)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 2 (2)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lip dry (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Dysuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 5 (5) | 3 (3) | 2 (2)
Hematuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 7 (7) | 6 (6) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 6 (6) | 7 (7) | 2 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 6 (6) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Onycholysis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 7 (7) | 0 (0) | 3 (3)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 9 (9) | 8 (8) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 11 (11) | 6 (6) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 10 (10) | 8 (8) | 3 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 5 (5) | 4 (4) | 3 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 6 (6) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 5 (5) | 2 (2) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 3 (3) | 3 (3) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (3) | 4 (4) | 15 (15) | 8 (8) | 9 (9)
Decreased appetite (Metabolism and nutrition disorders) | 6 (6) | 2 (2) | 14 (14) | 13 (13) | 6 (6)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 6 (6) | 8 (8) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 3 (3) | 7 (7) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 4 (4) | 6 (6) | 5 (5)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 3 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Bacteriuria (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localized infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Rocky mountain spotted fever (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1) | 8 (8) | 4 (4) | 3 (3)
Vaginitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Enterococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Impetigo (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes